CLINICAL TRIAL: NCT00286260
Title: Double-blind, Randomised, Placebo-controlled Trial of the Effect of Levetiracetam on Painful Polyneuropathy
Brief Title: Levetiracetam for Painful Polyneuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Professor Søren H. Sindrup, Odense University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: keppra2
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2006-01

CONDITIONS: Painful Polyneuropathy
Keywords: polyneuropathy; neuropathic pain; levetiracetam
MeSH Terms: conditions — Polyneuropathies; Neuralgia | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: levetiracetam — Levetiracetam tablet 500 mg, daily dose titrated to 3000 mg, 6 weeks

SUMMARY:
Polyneuropathy of different etiologies is often associated with pain. The standard treatment of this pain is anticonvulsants or antidepressants, but none of these treatment are effective or tolerable for all patients. Levetiracetam is a newer anticonvulsant and it is the hypothesis is that it could relieve neuropathic pain in polyneuropathy. This is a randomised, double-blind, placebo-controlled, cross-over trial on the effect of levetiracetam 3.000 mg/day on pain in polyneuropathy

ELIGIBILITY:
Inclusion Criteria:

* age 20 to 0 years
* painful symptoms of polyneuropathy for at least 6 months
* confirmed diagnosis of polyneuropathy
* baseline pain score of 4 or more (0 to 10 point scale)
* pain at least 4 days a week
* adequate anticonceptive treatment for women with childbearing potential
* informed consent

Exclusion Criteria:

* other cause of pain
* previous allergic reactions towards levetiracetam
* known adverse drug reactions on levetiracetam
* pregnancy
* severe disease
* inability to follow study protocol
* treatment with antidepressants, other anticonvulsants or opioids

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Pain relief rated on a 0 to 10 point numeric rating scale (median value for last treatment week in each period) | Daily

SECONDARY OUTCOMES:
Pain rated on 0 to 10 point numeric rating scales | Daily
Pain subtypes rated on 0 to 10 point numeric rating scales | Daily
Bruch-evoked pain | Baseline and end of each treament period
Pin-prick evoked pain | Baseline and end of each treatment period
Cold evoked pain | Baseline and end of each treatment period
Health related quality of life(SF-36) | Baseline and end of each treatment period
Pain related sleep disturbance | Daily
Use of escape medication | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Søren H Sindrup, Professor, Study Chair — Department of Neurology, Odense Unviersity Hospital
Locations (1):
- Department of Neurology, Odense University Hospital, Odense C, Denmark